CLINICAL TRIAL: NCT05766618
Title: The Effect of Multiple Injections of Platelets Rich Fibrin (i-PRF) on The Rate of Canine Retraction A Split-mouth: A Randomized Controlled Trial
Brief Title: The Effect of Multiple Injections of (PRF) on The Rate of Canine Retraction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mohamed Elmoghazy Alkhawaga, Doctor: Mohamed Mamdouh Mohamed Elmoghazy Alkhawaga, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I-PRF in orthodontics
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Platelet-Rich Fibrin; Acceleration; Orthodontics
Keywords: injectable platelets rich fibrin
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Intervention Model Description: This study is a split-mouth randomized, controlled single-center superiority trial, with two parallel groups with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injection site (Experimental): it is the arm where the patients will receive the PRF injection intraligamentally in distobuccal, and distopalatal areas of the distal surface of the canine also submucosal injection will be given buccally and palatially (0.25mm) for each side in either the right or left side of the arch.
  Interventions: Procedure: Injectable platelet rich fibrin (i-PRF): in acceleration of orthodontic tooth movement
- control site (No Intervention): it is the arm where the patients will not receive any injection with the same method of retraction as the intervention side.

INTERVENTIONS:
Procedure: Injectable platelet rich fibrin (i-PRF): in acceleration of orthodontic tooth movement — Preparatory phase
  * Space closure will be done on a 17x25 stainless steel wire
  * Both molars will be indirectly anchored to the miniscrew
  * Extend closing coil spring of suitable length from the canine hock to the first molar hock for retraction.
  * Apply a force of 150gm for each side. The force is measured by a force gauge and activated each visit to keep it constant all over the retraction phase. PRF Injection protocol
  * The First injection will be 3 weeks before extraction
  * By the end of the fourth week the patients will be referred for pre-intervention records. Upper arch CBCT will be obtained to take preintervention measurements of the alveolar bone.
  * At the time of canine retraction patient will receive another injection immediately and an alginate impression will be taken
  * follow up every month and injection will be repeated month after month with an observational period of 5 months.
  Other Names: The effect of autologous platelet concentrates on orthodontic tooth movement
  Arms: injection site

SUMMARY:
this clinical trial aims to prove that multiple injections will produce a steady rate of acceleration of orthodontic tooth movement.

DETAILED DESCRIPTION:
Platelet-rich fibrin injection is a second-generation platelet concentrate, prepared from centrifuged blood which is a rich source of platelets, stem cells, and growth factors seven times greater than that released by platelet-rich plasma. It is a simplified procedure with no biochemical manipulation of blood, free from anticoagulants which are known to inhibit wound healing or any gelling agent, and easily usable with a low rate of mistakes during the preparation procedure.

A variety of growth factors are released by PRF such as platelet-derived growth factor (PDGF), transforming growth factor β (TGF-β), and vascular endothelial growth factor (VEGF), which play a crucial role in angiogenesis, collagen synthesis, and bone regeneration.

Treatment with extraction especially in adult patients may take a longer time due to reported increase in bone density and lower bone regenerative rate. Also, the retraction process to close extraction spaces most of the time is accompanied by bone loss and root resorption as reported in the previous studies. i-PRF can accelerate tooth movement, in addition, prevent tooth retraction undesirable side effects.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* Full set of permanent dentition (excluding third molars).
* Good oral hygiene
* protrusion cases that require extraction of premolars (Bimaxillary protrusion or class II div 1)

Exclusion Criteria:

* History of previous orthodontic treatment.
* Systemic disease or drugs affecting tooth movement.
* Smokers
* Poor oral health that precludes orthodontic treatment (presence of caries, active white spots, or periodontal diseases)
* Severe crowding cases with ectopic erupted canines

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of canine retraction. | 5 months
  Rate of orthodontic tooth movement will be measured by calculating the difference in the canine position in mm throughout digital superimposition of consecutive digital models that will be made every four weeks.

SECONDARY OUTCOMES:
1. Assess bone level between intervention and control side. | bone level will be measured at the beginning of the study (T1) and by the fifth month of the study (T5)
  1. bone level between intervention and control side will be assessed through pre and post retraction CBCT for the upper arch.

OTHER OUTCOMES:
Assess Periodontal health at the injection side. | 5 months
  2. Assess Periodontal health on the injection side through periodontal charting mainly propping depth.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Alkhawaga, BDS, Principal Investigator — Cairo University; Fady Fahim, phD, Study Director — Cairo University; Sally Magdy, phD, Study Chair — Cairo University
Locations (1):
- Vice president of graduate studies of Cairo University, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Result] Aboalnaga AA, Salah Fayed MM, El-Ashmawi NA, Soliman SA. Effect of micro-osteoperforation on the rate of canine retraction: a split-mouth randomized controlled trial. Prog Orthod. 2019 Jun 3;20(1):21. doi: 10.1186/s40510-019-0274-0. PMID 31155698
- [Result] Huang H, Williams RC, Kyrkanides S. Accelerated orthodontic tooth movement: molecular mechanisms. Am J Orthod Dentofacial Orthop. 2014 Nov;146(5):620-32. doi: 10.1016/j.ajodo.2014.07.007. Epub 2014 Oct 28. PMID 25439213
- [Result] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- [Result] El-Timamy A, El Sharaby F, Eid F, El Dakroury A, Mostafa Y, Shaker O. Effect of platelet-rich plasma on the rate of orthodontic tooth movement. Angle Orthod. 2020 May 1;90(3):354-361. doi: 10.2319/072119-483.1. PMID 33378433
- [Result] Erdur EA, Karakasli K, Oncu E, Ozturk B, Hakki S. Effect of injectable platelet-rich fibrin (i-PRF) on the rate of tooth movement. Angle Orthod. 2021 May 1;91(3):285-292. doi: 10.2319/060320-508.1. PMID 33459765
- [Result] KINGSLEY CS. Blood coagulation; evidence of an antagonist to factor VI in platelet-rich human plasma. Nature. 1954 Apr 17;173(4407):723-4. doi: 10.1038/173723a0. No abstract available. PMID 13165629
- [Result] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Result] He L, Lin Y, Hu X, Zhang Y, Wu H. A comparative study of platelet-rich fibrin (PRF) and platelet-rich plasma (PRP) on the effect of proliferation and differentiation of rat osteoblasts in vitro. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Nov;108(5):707-13. doi: 10.1016/j.tripleo.2009.06.044. PMID 19836723
- [Result] Dohan Ehrenfest DM, Del Corso M, Diss A, Mouhyi J, Charrier JB. Three-dimensional architecture and cell composition of a Choukroun's platelet-rich fibrin clot and membrane. J Periodontol. 2010 Apr;81(4):546-55. doi: 10.1902/jop.2009.090531. PMID 20373539
- [Result] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Result] Del Corso M, Vervelle A, Simonpieri A, Jimbo R, Inchingolo F, Sammartino G, Dohan Ehrenfest DM. Current knowledge and perspectives for the use of platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) in oral and maxillofacial surgery part 1: Periodontal and dentoalveolar surgery. Curr Pharm Biotechnol. 2012 Jun;13(7):1207-30. doi: 10.2174/138920112800624391. PMID 21740371
- [Result] Reichert C, Kutschera E, Plotz C, Scharf S, Golz L, Fimmers R, Fuhrmann C, Wahl G, Braumann B, Jager A. Incidence and severity of gingival invaginations associated with early versus late initiation of orthodontic space closure after tooth extraction : A multicenter pilot and randomized controlled trial. J Orofac Orthop. 2017 Sep;78(5):415-425. doi: 10.1007/s00056-017-0098-9. Epub 2017 Jun 28. PMID 28660421
- [Result] Farshidfar N, Amiri MA, Firoozi P, Hamedani S, Ajami S, Tayebi L. The adjunctive effect of autologous platelet concentrates on orthodontic tooth movement: A systematic review and meta-analysis of current randomized controlled trials. Int Orthod. 2022 Mar;20(1):100596. doi: 10.1016/j.ortho.2021.10.004. Epub 2021 Dec 2. PMID 34866025
- [Result] Sivarajan S, Ringgingon LP, Fayed MMS, Wey MC. The effect of micro-osteoperforations on the rate of orthodontic tooth movement: A systematic review and meta-analysis. Am J Orthod Dentofacial Orthop. 2020 Mar;157(3):290-304. doi: 10.1016/j.ajodo.2019.10.009. PMID 32115107
- [Result] Mheissen S, Khan H, Alsafadi AS, Almuzian M. The effectiveness of surgical adjunctive procedures in the acceleration of orthodontic tooth movement: A systematic review of systematic reviews and meta-analysis. J Orthod. 2021 Jun;48(2):156-171. doi: 10.1177/1465312520988735. Epub 2021 Feb 5. PMID 33546565
- [Result] Alfailany DT, Hajeer MY, Aljabban O, Mahaini L. The Effectiveness of Repetition or Multiplicity of Different Surgical and Non-Surgical Procedures Compared to a Single Procedure Application in Accelerating Orthodontic Tooth Movement: A Systematic Review and Meta-Analysis. Cureus. 2022 Mar 12;14(3):e23105. doi: 10.7759/cureus.23105. eCollection 2022 Mar. PMID 35296053
- [Result] Figueiredo DS, Houara RG, Pinto LM, Diniz AR, de Araujo VE, Thabane L, Soares RV, Oliveira DD. Effects of piezocision in orthodontic tooth movement: A systematic review of comparative studies. J Clin Exp Dent. 2019 Nov 1;11(11):e1078-e1092. doi: 10.4317/jced.56328. eCollection 2019 Nov. PMID 31700581
- [Result] Elmotaleb MAA, Elnamrawy MM, Sharaby F, Elbeialy AR, ElDakroury A. Effectiveness of using a Vibrating Device in Accelerating Orthodontic Tooth Movement: A Systematic Review and Meta-Analysis. J Int Soc Prev Community Dent. 2019 Jan-Feb;9(1):5-12. doi: 10.4103/jispcd.JISPCD_311_18. Epub 2019 Feb 14. PMID 30923687
- [Result] Bakdach WMM, Hadad R. Effectiveness of low-level laser therapy in accelerating the orthodontic tooth movement: A systematic review and meta-analysis. Dent Med Probl. 2020 Jan-Mar;57(1):73-94. doi: 10.17219/dmp/112446. PMID 32314880
- [Result] Imani MM, Golshah A, Safari-Faramani R, Sadeghi M. Effect of Low-level Laser Therapy on Orthodontic Movement of Human Canine: a Systematic Review and Meta-analysis of Randomized Clinical Trials. Acta Inform Med. 2018 Jun;26(2):139-143. doi: 10.5455/aim.2018.26.139-143. PMID 30061788
- [Result] Arqub SA, Gandhi V, Iverson MG, Ahmed M, Kuo CL, Mu J, Dutra E, Uribe F. The effect of the local administration of biological substances on the rate of orthodontic tooth movement: a systematic review of human studies. Prog Orthod. 2021 Feb 1;22(1):5. doi: 10.1186/s40510-021-00349-5. PMID 33523325
- [Result] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995
- [Result] Gollapudi M, Bajaj P, Oza RR. Injectable Platelet-Rich Fibrin - A Revolution in Periodontal Regeneration. Cureus. 2022 Aug 31;14(8):e28647. doi: 10.7759/cureus.28647. eCollection 2022 Aug. PMID 36196318
- [Result] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Three-dimensional evaluation of the effects of injectable platelet rich fibrin (i-PRF) on alveolar bone and root length during orthodontic treatment: a randomized split mouth trial. BMC Oral Health. 2021 Mar 2;21(1):92. doi: 10.1186/s12903-021-01456-9. PMID 33653326
- [Result] Miron RJ, Fujioka-Kobayashi M, Bishara M, Zhang Y, Hernandez M, Choukroun J. Platelet-Rich Fibrin and Soft Tissue Wound Healing: A Systematic Review. Tissue Eng Part B Rev. 2017 Feb;23(1):83-99. doi: 10.1089/ten.TEB.2016.0233. Epub 2016 Oct 10. PMID 27672729
- [Result] Cagli Karci I, Baka ZM. Assessment of the effects of local platelet-rich fibrin injection and piezocision on orthodontic tooth movement during canine distalization. Am J Orthod Dentofacial Orthop. 2021 Jul;160(1):29-40. doi: 10.1016/j.ajodo.2020.03.029. Epub 2021 May 4. PMID 33962809
- [Result] Gupta P, Bhagyalakshmi A, Avinash BS, Prashant A, Raghunath N. Evaluation of injectable platelet-rich fibrin effect on the rate of canine retraction and alkaline phosphatase levels: An in-vivo study. Am J Orthod Dentofacial Orthop. 2022 Nov;162(5):735-743. doi: 10.1016/j.ajodo.2021.07.019. Epub 2022 Aug 23. PMID 36008239
- [Result] Mheissen S, Daraqel B, Alzoubi EE, Khan H. Effectiveness of platelet-rich concentrates on the rate of orthodontic tooth movement: a systematic review and meta-analysis. Eur J Orthod. 2023 Mar 31;45(2):196-207. doi: 10.1093/ejo/cjac049. PMID 36056906
- [Result] Choukroun J, Ghanaati S. Reduction of relative centrifugation force within injectable platelet-rich-fibrin (PRF) concentrates advances patients' own inflammatory cells, platelets and growth factors: the first introduction to the low speed centrifugation concept. Eur J Trauma Emerg Surg. 2018 Feb;44(1):87-95. doi: 10.1007/s00068-017-0767-9. Epub 2017 Mar 10. PMID 28283682
- [Result] Song D, Shujaat S, de Faria Vasconcelos K, Huang Y, Politis C, Lambrichts I, Jacobs R. Diagnostic accuracy of CBCT versus intraoral imaging for assessment of peri-implant bone defects. BMC Med Imaging. 2021 Feb 10;21(1):23. doi: 10.1186/s12880-021-00557-9. PMID 33568085
- [Result] Adarsh K, Sharma P, Juneja A. Accuracy and reliability of tooth length measurements on conventional and CBCT images: An in vitro comparative study. J Orthod Sci. 2018 Sep 6;7:17. doi: 10.4103/jos.JOS_21_18. eCollection 2018. PMID 30271762